CLINICAL TRIAL: NCT06506383
Title: Geographical Variations and Predictors of Coronary Artery Disease Mortality in Turkiye: An Environmental and Behavioral Analysis
Brief Title: Coronary Artery Disease Mortality in Turkiye
Status: Completed | Type: Observational
Sponsor: Medipol University (Other)
Responsible Party: Principal Investigator, Mehmet Kocak, Professor and Chair of Biostatistics, Medipol University
Other Study IDs: CAD001
Record Dates: First submitted 2024-07-11; First posted 2024-07-17 (Actual); Last update posted 2024-07-17 (Actual); Status verified 2024-07

CONDITIONS: Coronary Artery Disease (CAD) Mortality
MeSH Terms: conditions — Coronary Artery Disease

STUDY DESIGN:
Observational Model: Ecologic or Community | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: No Intervention as this is an ecological study — No Intervention as this is an ecological study

SUMMARY:
This study aims to analyze the geographical variations and identify key environmental and behavioral predictors of coronary artery disease (CAD) mortality in Turkiye.

DETAILED DESCRIPTION:
A 10-year longitudinal province-level data was used to identify change trajectories of CAD mortality. . Environmental determinants (such as air quality and climatic conditions) and behavioral factors of alcohol consumption and smoking were examined for their association with CAD mortality change trajectories using Ordinal Logistic Regression models.

ELIGIBILITY:
Inclusion Criteria:

* All citizens in a given province

Exclusion Criteria:

* None

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: The study population includes all citizens in each of the 81 provinces of Turkiye
Sampling Method: Non-Probability Sample
Enrollment: 81 (Actual)
Dates: Start 2020-01-01 (Actual); Primary Completion 2022-12-31 (Actual); Study Completion 2023-06-30 (Actual)

PRIMARY OUTCOMES:
CAD Mortality | 2010-2019
  coronary artery disease (CAD) mortality per 100,000 population

CONTACTS AND LOCATIONS:
Locations (1):
- Istanbul Medipol University, Beykoz, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
These are national mortality data and we cannot share it